CLINICAL TRIAL: NCT00314262
Title: Phase I/II Study of Chemoprevention With Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor Erlotinib (OSI-774, Tarceva) and Cyclooxygenase-2 (COX-2) Inhibitor (Celecoxib) in Premalignant Lesions of Head and Neck of Former Smokers
Brief Title: Phase I/II Study of Chemoprevention With EGFR and COX-2 Inhibitor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Dong Shin, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00024922
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Precancerous Conditions
Keywords: Skin Lesions; Premalignant Lesion
MeSH Terms: conditions — Precancerous Conditions | interventions — Erlotinib Hydrochloride; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib & Celecoxib (Experimental)
  Interventions: Drug: Erlotinib & Celecoxib

INTERVENTIONS:
Drug: Erlotinib & Celecoxib — Erlotinib given orally, once daily (dose escalation from 50 mg, 75 mg, or 100 mg) continuously for 6 months in the phase I portion.
  Celecoxib given 400 mg orally BID continuously for 6 months.
  Other Names: OSI-774, Tarceva

SUMMARY:
Evaluate effect on cells and patient response to study medications, assess side effects of these medications, and evaluate chemicals in cells that may tell how the drug works, before, and after receiving the study medications.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect on cells and patient response to study medications, assess the side effects of these medications, and to evaluate chemicals in the cells that may tell how the drug works, before, and after receiving the study medications.

Approximately 61 patients will participate at Emory Winship Cancer Institute and Emory Crawford W. Long Hospital in Atlanta, Georgia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have premalignant lesions.
* Lesion sites include oral cavity, oropharynx, and larynx.
* Must have at least a >20 pack-year history of smoking.
* Must have a Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status of 0-1.
* Participants must be 18 years of age or older.
* No contraindications for laryngoscopy and biopsy.
* Adequate liver function.
* Must have hemoglobin and hematocrit levels at or above the lower limit of the normal range.
* Participants must have prothrombin time (PT)/partial thromboplastin time (PTT) levels at or above the lower limit of the normal range.
* Women of child-bearing potential must have a negative serum pregnancy test within 72 hours of receiving treatment.
* Must be able to swallow the oral dose of erlotinib and celecoxib.
* Participants must be disease free.
* Final eligibility will be determined by the health professionals conducting the trial.

Exclusion Criteria:

* Participants with acute intercurrent illness or those who had surgery within the preceding 4 weeks unless they have fully recovered.
* History of previous malignancies unless the cancer was stage I or II and rendered free of disease more than 1 year.
* Pregnant or breast feeding.
* Not practicing adequate contraception if the participants are of child bearing potential.
* Female patients who have a positive pregnancy test.
* History or recent myocardial infarction.
* Hypertension not adequately controlled by medication.
* Documented history of coagulopathy.
* Documented history of congestive heart failure (CHF) greater than New York Heart Association (NYHA) Grade II.
* Participants who were taking COX-2 inhibitors or EGFR tyrosine kinase inhibitors within 3 months of study entry.
* Documented history or interstitial lung disease.
* Known connective tissue disease.
* History of nonsteroidal antiinflammatory drug (NSAID)-induced ulcers or those who are at risk for a GI ulcer.
* Participated in a clinical trial of an investigational drug within 12 months prior to enrollment.
* Final eligibility will be determined by the health professionals conducting the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Shin, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Background] Shin DM, Zhang H, Saba NF, Chen AY, Nannapaneni S, Amin AR, Muller S, Lewis M, Sica G, Kono S, Brandes JC, Grist WJ, Moreno-Williams R, Beitler JJ, Thomas SM, Chen Z, Shin HJ, Grandis JR, Khuri FR, Chen ZG. Chemoprevention of head and neck cancer by simultaneous blocking of epidermal growth factor receptor and cyclooxygenase-2 signaling pathways: preclinical and clinical studies. Clin Cancer Res. 2013 Mar 1;19(5):1244-56. doi: 10.1158/1078-0432.CCR-12-3149. Epub 2013 Feb 19. PMID 23422093
- [Result] Saba NF, Hurwitz SJ, Kono SA, Yang CS, Zhao Y, Chen Z, Sica G, Muller S, Moreno-Williams R, Lewis M, Grist W, Chen AY, Moore CE, Owonikoko TK, Ramalingam S, Beitler JJ, Nannapaneni S, Shin HJ, Grandis JR, Khuri FR, Chen ZG, Shin DM. Chemoprevention of head and neck cancer with celecoxib and erlotinib: results of a phase ib and pharmacokinetic study. Cancer Prev Res (Phila). 2014 Mar;7(3):283-91. doi: 10.1158/1940-6207.CAPR-13-0215. Epub 2013 Oct 3. PMID 24085777

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 24, 2006, and June 28, 2012, 36 subjects with documented premalignant lesions, including mild (mild-D), moderate, or severe oral leukoplakia, and carcinoma in situ (CIS) were screened. Lesion sites included oral cavity oropharynx, and the larynx.
Pre-assignment Details: Seventeen subjects were enrolled on the study, 3 of whom withdrew consent (one male of 69 years of age, and two females of 43 and 42 years of age). Two patients who signed informed consent were deemed to be screen failures, one secondary to prior history of oral squamous cell carcinoma and the other secondary to a history of cardiac arrhythmias.
Period: Overall Study
Arm/Group | Erlotinib & Celecoxib
Started | 12
Completed | 7
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib & Celecoxib
Number analyzed (Participants) | 12
Age, Customized [Number; unit: participants]
  40-49 years old | 4
  50-59 years old | 2
  60-69 years old | 4
  70-79 years old | 1
  80-89 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation and Toxicity: Toxicities Including Grades 1 to 4
Description: Participants received a fixed dose of celecoxib 400 mg orally BID continuously for 6 months. Erlotinib was dose escalated at 3 dose levels of 50, 75, and 100 mg orally every day for 6 months. Dose escalation followed a standard 3+3 escalation design.
Time Frame: 12 months from time of enrollment
Measure: Number; unit: participants
Arm/Group | Erlotinib & Celecoxib
Number analyzed (Participants) | 7
participants
  Abdominal cramping, Grade 1 | 2
  Alopecia, Grade 1 | 2
  Anemia, Grade 1 | 2
  Anemia, Grade 2 | 1
  Anxiety, Grade 1 | 2
  Decreased protein, Grade 1 | 2
  Leukopenia, Grade 1 | 1
  Leukopenia, Grade 2 | 1
  Depression, Grade 1 | 3
  Diarrhea, Grade 1 | 5
  Dry eyes, Grade 1 | 4
  Dry skin, Grade 1 | 6
  Elevated LDH, Grade 1 | 3
  Elevated serum creatinine, Grade 1 | 4
  Elevated serum creatinine, Grade 2 | 1
  Elevated alkaline phosphatase, Grade 1 | 3
  Elevated ALT, Grade 1 | 5
  Elevated AST, Grade 4 | 4
  Fatigue, Grade 1 | 6
  Hyperbilirubinemia, Grade 1 | 2
  Hypercholesterolemia, Grade 1 | 2
  Hyperglycemia, Grade 1 | 7
  Hyperglycemia, Grade 2 | 2
  Hypoalbuminemia, Grade 1 | 3
  Hypoalbuminemia, Grade 2 | 1
  Hypocalcemia, Grade 1 | 4
  Hypoglycemia, Grade 1 | 1
  Hypoglycemia, Grade 2 | 1
  Hypokalemia, Grade 1 | 2
  Hyponatremia, Grade 1 | 3
  Mouth sores, Grade 1 | 9
  Mouth sores, Grade 2 | 3
  Mucositis, Grade 1 | 3
  Mucositis, Grade 3 | 1
  Nausea, Grade 1 | 4
  Neuropathy, Grade 1 | 3
  Pruritis, Grade 1 | 2
  Rash, Grade 1 | 8
  Rash, Grade 3 | 2
  Shortness of breath, Grade 1 | 3
  Strep throat, Grade 2 | 1
  Urosepsis, Grade 3 | 1
  Vomiting, Grade 1 | 2

2. Primary Outcome: Clinical Outcome: Documented Progression
Description: Response evaluation was based on pathologic examination of the degree of dysplasia observed and recorded by an expert head and neck pathologist. Pathologic complete response was defined as complete disappearance of dysplasia from the epithelium. Pathologic partial response was defined as improvement of dysplasia by at least one degree (i.e., severe dysplasia becomes moderate dysplasia). Pathologic minor response or stable disease was defined as minor focal improvement without change of degree of dysplasia (i.e., focal improvement from moderate to mild dysplasia with still moderate dysplasia overall) or no pathologic changes after treatment. Pathologic progressive disease was defined as worsening by at least one degree of dysplasia (i.e., mild to moderate dysplasia) or development of invasive cancer on or following treatment.
Time Frame: 12 months from time of enrollment
Measure: Number; unit: participants
Arm/Group | Erlotinib & Celecoxib
Number analyzed (Participants) | 7
participants
  Complete remission (CR) | 3
  Partial remission (PR) | 1
  Progressive disease (PD) | 1
  Stable disease (SDi) | 2

3. Primary Outcome: Clinical Outcome: Progression to a Higher-grade Dysplasia or Carcinoma
Description: as for outcome 2
Time Frame: Up to 55 months from initiation of therapy. Median duration of follow-up was 36 months.
Measure: Number; unit: participants
Arm/Group | Erlotinib & Celecoxib
Number analyzed (Participants) | 7
participants
  Stage I invasive carcinoma | 1
  Stage II oral cavity carcinoma | 1
  Invasive squamous cell carcinoma | 1
  Recurrent moderate dysplasia | 1
  Recurrent severe dysplasia | 1
  Recurrent high-grade dysplasia | 1
  Complete remission | 1

ADVERSE EVENTS:
Arm/Group | Erlotinib & Celecoxib
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib & Celecoxib (N=12)
Rash (Grade 3) (Skin and subcutaneous tissue disorders) | 1
Mucositis (Grade 3) (Gastrointestinal disorders) | 1
Urosepsis (Grade 3) (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib & Celecoxib (N=12)
Abdominal cramping (Grade 1) (Gastrointestinal disorders) | 2
Alopecia (Grade 1) (Renal and urinary disorders) | 2
Anemia (Grade 1) (Blood and lymphatic system disorders) | 2
Anemia (Grade 2) (Blood and lymphatic system disorders) | 1
Anxiety (Grade 1) (Psychiatric disorders) | 2
Decreased protein (Grade 1) (Blood and lymphatic system disorders) | 2
Leukopenia (Grade 1) (Immune system disorders) | 1
Leukopenia (Grade 2) (Immune system disorders) | 1
Depression (Grade 1) (Psychiatric disorders) | 3
Diarrhea (Grade 1) (Gastrointestinal disorders) | 5
Dry Eyes (Grade 1) (Eye disorders) | 4
Dry Skin (Grade 1) (Skin and subcutaneous tissue disorders) | 6
Elevated Lactate Dehydrogenase (Grade 1) (Blood and lymphatic system disorders) | 3
Elevated Serum Creatinine (Grade 1) (Renal and urinary disorders) | 4
Elevated Alkaline Phosphatase (Grade 1) (Blood and lymphatic system disorders) | 3
Elevated Alanine Aminotransferase (Grade 1) (Blood and lymphatic system disorders) | 5
Elevated Aspartate Aminotransferase (Grade 1) (Blood and lymphatic system disorders) | 4
Fatigue (Grade 1) (General disorders) | 6
Hyperbilirubinemia (Grade 1) (Blood and lymphatic system disorders) | 2
Hypercholesterolemia (Grade 2) (Blood and lymphatic system disorders) | 2
Hyperglycemia (Grade 1) (Blood and lymphatic system disorders) | 7
Hyperglycemia (Grade 2) (Blood and lymphatic system disorders) | 2
Hypoalbuminemia (Grade 1) (Blood and lymphatic system disorders) | 3
Hypoalbuminemia (Grade 2) (Blood and lymphatic system disorders) | 1
Hypocalcemia (Grade 1) (Blood and lymphatic system disorders) | 4
Hypoglycemia (Grade 1) (Blood and lymphatic system disorders) | 1
Hypoglycemia (Grade 2) (Blood and lymphatic system disorders) | 1
Hypokalemia (Grade 1) (Blood and lymphatic system disorders) | 2
Hyponatremia (Grade 1) (Blood and lymphatic system disorders) | 3
Mouth Sores (Grade 1) (Skin and subcutaneous tissue disorders) | 9
Mouth Sores (Grade 2) (Skin and subcutaneous tissue disorders) | 3
Mucositis (Grade 1) (Gastrointestinal disorders) | 3
Nausea (Grade 1) (General disorders) | 4
Neuropathy (Grade 1) (Nervous system disorders) | 3
Pruritis (Grade 1) (Skin and subcutaneous tissue disorders) | 2
Rash (Grade 1) (Skin and subcutaneous tissue disorders) | 8
Shortness of Breath (Grade 1) (General disorders) | 3
Strep Throat (Grade 2) (Infections and infestations) | 1
Vomiting (Grade 1) (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
One limitation is the small number of patients who were evaluable for response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes